CLINICAL TRIAL: NCT02131142
Title: To Collect Additional Safety and Effectiveness Data for the Biosensors BioFreedom™ BA9 Drug Coated Coronary Stent in Patients With Native, de Novo Coronary Artery Disease
Brief Title: BioFreedom US IDE Feasibility Trial
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Biosensors Europe SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14US01
Record Dates: First submitted 2014-05-05; First posted 2014-05-06 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Ischemic Heart Disease; Stable Angina; Unstable Angina; Silent Ischemia
Keywords: ischemic heart disease; CAD
MeSH Terms: conditions — Myocardial Ischemia; Angina, Stable; Angina, Unstable

ARMS (1):
- BioFreedom (Experimental)
  Interventions: Device: BioFreedom drug coated coronary stent

INTERVENTIONS:
Device: BioFreedom drug coated coronary stent — Placement of a BioFreedom drug coated stent in a narrow coronary artery

SUMMARY:
The purpose of this study is to collect additional safety and effectiveness data for on the Biosensors BioFreedom™ BA9 Drug Coated Coronary Stent in patients with native, de novo coronary artery disease.

DETAILED DESCRIPTION:
This is a multi-center prospective trial of 100 patients at up to 15 centers. The study population will consist of patients preventing with symptomatic ischemic heart disease due to de novo stenotic lesion(s) in native coronary artery(ies) with reference vessel diameter between 2.25 mm and 4.0 mm.

The primary safety endpoint for this clinical trial is the occurrence of major adverse cardiac events (MACE) defined as the composite of cardiac death, myocardial infarction, target lesion revascularization and academic research consortium (ARC) definite stent thrombosis within 9 months following the implantation.

The primary effectiveness endpoint for this trial is in-stent late lumen loss at 9 months as compared to historical control

ELIGIBILITY:
Inclusion Criteria:

* Individual is ≥ 18 years of age
* Individual must have clinical evidence if ischemic heart disease, stable or unstable angina, silent ischemia, or a positive functional study;
* Individual must be an acceptable candidate for percutaneous coronary intervention (PCI), stenting, and emergent coronary artery bypass graft (CABG) surgery
* Individual is competent and willing to provide informed consent to participate in the trial

Exclusion Criteria:

* A known hypersensitivity or contraindication to aspirin, heparin, clopidogrel, or a sensitivity to contrast media that cannot be adequately pre-medicated;
* History or known allergic reaction or significant sensitivity to drugs similar to BA9;
* A platelet count < 100,000 cells/mm3 or > 700,000 cells/mm3, or a WBC < 3,000 cells/mm3;
* A creatinine level > 2.5 mg/dL;
* Evidence of an acute myocardial infarction with 72 hours of the intended stenting (defined as: Q wave or non-Q wave myocardial infarction having a Troponin either I or T pre-procedure elevated above the Institution's upper limit of normal);
* Previous or planned PCI of any vessel within 30 days pre or post procedure;
* Patient unable to take clopidogrel for 3 months or patient who have comorbidities that would prohibit the cessation of clopidogrel at 3 months;
* Planned adjunctive treatment during the intended stenting (eg balloon valvuloplasty, percutaneous endovascular intervention, etc)
* During the intended or index procedure the target lesion(s) requires treatment with a device other than a plain old balloon prior to stent placement (such as, but not limited to, cutting balloon, directional atherectomy, excimer laser, rotational atherectomy, thrombectomy, etc);
* History of documented prior stroke within 6 months of the intended procedure;
* Active peptic ulcer or upper gastrointestinal bleeding documented within the prior 6 months;
* History of active bleeding diathesis or coagulopathy or will refuse blood transfusion;
* Individual is pregnant, nursing or planning to be pregnant;
* Any previous or planned treatment of the target vessel(s) with anti-restenotic therapies including, but not limited to brachytherapy;
* Concurrent medical condition with a life expectancy of less than 12 months or individual has any serious medical condition, which in the opinion of the investigator, may adversely affect the safety and/or effectiveness of the participant or the study;
* Individual is currently enrolled in another investigational drug or device trial. If, however, if investigational trial device or drug becomes commercially available, these trials are not considered investigational;
* Previous ACS within 9 months of pre or post procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2014-08; Primary Completion 2015-08 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Safety of the BioFreedom stent | 9 month
  The occurrence of major adverse cardiac events (MACE) defined as the composite of cardiac death, myocardial infarction, target lesion revascularization and academic research consortium (ARC) definite stent thrombosis
Efficacy of the BioFreedom stent | 9 month
  Stent late lumen loss at 9 months as compared to historical control

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Baptist Cardiac & Vascular Institute, Miami, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Jewish Hospital and Saint Mary's Healthcare, Louisville, Kentucky
  - MedStar Union Memorial Hospital, Baltimore, Maryland
  - MedStar Southern Maryland Hospital Center, Clinton, Maryland
  - Cardiac & Vascular Research Center of Northern Michigan, Petoskey, Michigan
  - Our Lady of Lourdes Medical Center, Voorhees Township, New Jersey
  - Columbia University Medical Center, New York, New York
  - NC Heart and Vascular Research-Rex Hospital, Raleigh, North Carolina
  - The Carl & Edyth Lindner Center for Research, Cincinnati, Ohio
  - Mercy St. Vincent Medical Center, Toledo, Ohio
  - Berks Cardiology, Wyomissing, Pennsylvania